CLINICAL TRIAL: NCT03470298
Title: Retrieval Endometrial Scratching Versus Mid-luteal Endometrial Scratching for Women Undergoing ICSI for Unexplained Infertility
Brief Title: Retrieval Versus Mid-luteal Endometrial Scratching (ES) for Intra Cytoplasmic Sperm Injection (ICSI)
Acronym: ICSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abd Elhady Zayed, Associate professor of Obstetrics &Gynecology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: R/16.11.11; ABC123 (Registry Identifier: Mansoura university)
Record Dates: First submitted 2018-03-07; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: ICSI
Keywords: Endometrial Scratching; Unexplained infertility; ICSI

STUDY DESIGN:
Intervention Model Description: The patients in study undergo endometrial scratch technique after being randomly assigned in to one of two groups . First group undergo ES just after finishing oocyte pick up and the other group undergo ES one week before starting COH. Manual Vacuum Aspiration (MVA) size 5 moved from below upwards with suction ,scratching anterior uterine wall then posterior then left lateral uterine wall then right lateral uterine wall and lastly funds.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mid luteal Endometrial Scratching (MLES) (Active Comparator): Making injury to endometrium by using Manual Vacuum Aspiration cannula size 5 . At this arm scratching done at mid luteal phase (day21) of the cycle before induction for ICSI
  Interventions: Procedure: Endometrial scratching
- Retrieval Endometrial Scratching (RES) (Active Comparator): Making injury to endometrium by using Manual Vacuum Aspiration cannula size 5 .Here scratching done at same day of ovum pick up of ICSI cycle the difference only between arm of MLES and RES only in the timing of scratching .
  Interventions: Procedure: Endometrial scratching

INTERVENTIONS:
Procedure: Endometrial scratching — The patients in study undergo endometrial scratch technique after being randomly assigned in to one of two groups . First group undergo oocyte pickup just after finishing oocyte pick up and the other group undergo oocyte pickup one week before starting COH.ManualVaccum Aspiration (MVA) size 5 moved from below upwards with suction ,scrachning anterior uterine wall then posterior then left lateral uterine wall then right lateral uterine wall and lastly fundus. All patients were prescribed vibramycine 100 mg twice daily for 3 days starting one day before procedure
  Other Names: Endometrial injury

SUMMARY:
ES is a procedure used to help embryos to implant more successfully after In-Vitro Fertilization (IVF) , ICSI in patients who had failed cycles in spite of transfer of good quality embryos. New researches and evidence suggests that scratching the uterine endometrium causes a repair reaction in patients may increase embryo implantation rate . In spit of the optimum timing of scratching not finally determined, the usual timing to perform ES is approximately one week before starting IVF, ICSI treatment . our study aims to compare other time of scratching which is the scratching at retrieval time.

DETAILED DESCRIPTION:
Endometrial scratching (ES) is a procedure used to help embryos to implant more successfully after In-Vitro Fertilization (IVF), ICSI in patients who had failed cycles in spite of transfer of good quality embryos. New researches and evidence suggests that scratching the uterine endometrium causes a repair reaction in patients may increase embryo implantation rate. The usual timing to perform ES is approximately one week before starting IVF, ICSI treatment.

Aim:

Comparing results of performing endometrial scratching one week before starting ICSI cycle treatment and at day of oocyte retrieval.

Material &Methods :

This is a prospective clinical trial, involving patients undergoing ICSI treatment at fertility care unite, Mansoura University Hospital and private fertility centers. The subjects were recruited from the period between January 2017 and June 2018. An informed consent obtained. Sample size was calculated using Graph Pad Inset soft were, version 3.01.Twenty four patient in each group were required to give the study a power of 80% and α of 0.05. Good responders were defined as the patients who had develop, at least four good-quality embryos grade 1 and 2 of Veeck's grading in the previous IVF cycle. Patients found eligible for the study were offered to undergo endometrial scratch-suction either in The usual timing to perform ES is approximately one week before starting IVF, ICSI treatment, the other at the time of oocyte retrieval, just after finishing oocyte pickup.

All patients were evaluated with basal (day 3) Follicle Stimulating Hormone( FSH), and antral follicle count of the cycle prior to the embryo transfer cycle. Each woman recruited in the study underwent the same Controlled Ovarian Stimulation (COH) protocol that she had undergone in the previous ICSI cycles, which included only, long mid luteal phase Gonadotroph in Releasing Hormone (GnRH) agonist suppression . Records of previous stimulation protocols and embryology details were reviewed. The patients in study undergo endometrial scratch technique after being randomly assigned in to one of two groups. First group undergo oocyte pickup just after finishing oocyte pick up and the other group undergo oocyte pickup one week before starting COH. Manual Vacuum Aspiration (MVA) size 5 moved from below upwards with suction scratching anterior uterine wall then posterior then left lateral uterine wall then right lateral uterine wall and lastly fundus. All patients were prescribed vibramycine 100 mg twice daily for 3 days starting one day before procedure. In the long protocol, patients were down regulated with 0.1 mg GnRH agonist for the period of 10 - 14 days following which the dose was reduced to 0.5 mg and continued till human chorionic gonadotrophine (hCG) . After confirming adequate down-regulation, FSH, in the dose ranging from 150 to 250 IU, was commenced. FSH was continued till ovulation triggering .Women were scheduled for oocyte retrieval when at least three follicles reached a size of 18 mm. Oocyte retrieval was performed by the trans vaginal route under ultrasound guidance, 34-hr after HCG trigger with 5000 -1000 IU, with the patient under conscious sedation. The morphology of each aspirated oocyte was noted after denudation with hyaluronidase . ICSI was performed for all patients .The embryos were classified according to Veeck's grading as follows:

Grade 1 - preembryos with blastomeres of equal size and no cytoplasmic fragmentation; Grade 2 - preembryos with blastomeres of equal size with cytoplasmic fragmentation equal to 15% of the total embryonic volume.

Grade 3 - uneven blastomeres with no fragmentation; Grade 4 - uneven blastomeres with gross fragmentation (≥20% fragments) . Grade 1 or 2 embryos were considered to be good-quality embryos. Embryo transfer was performed with a Wallace® catheter (Smith Medical International Ltd., Hythe, Kent, UK) on day 3 a traumatically under ultrasound guidance by a senior consultant. we transfer up to three good-quality embryos. β-hCG was determined 2 weeks after the embryo transfer.

Statistical analysis All statistical analyses using SPSS for windows version 17.0 (SPSS, Chicago, IL). Continuous data were expressed as mean ±SD and compared between the two groups using independent Student's t test. Categorical data were expressed in number and percent and compared using the χ2 test. The 95 % confidence intervals (CI) for the difference in means were calculated. Statistical significance was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one previous failed ICSI cycles, Good responders in the previous ICSI cycle and Less than or equal to 35 years

Exclusion Criteria:. We excluded patients with; Presence of intramural fibroid distorting the endometrial cavity/sub mucous myoma/a Sherman's syndrome, Presence of son graphically detected hydrosalpinx, Patient age more than 35 years

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | about 9 months
  delivery of a fetus after passing medico legal viability

SECONDARY OUTCOMES:
implantation rate | 2 weeks after embryo transfer
  positive pregnancy test
Clinical pregnancy rate | 4 weeks after embryo transfer
  Appearance of gestational sac by ultrasound with fetal pole and cardiac pulsation

CONTACTS AND LOCATIONS:
Overall Officials: Abdelhady A Zayed, Ass. prof., Principal Investigator — Mansoura university hospital ,Mansoura,Dakahlia,Egypt
Locations (1):
- Fertility care unite,Mansoura university hospital., Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet decided if individual participant data will be available or not except after completion of study and counseling all persons sharing in the study .

REFERENCES:
- [Background] Barash A, Dekel N, Fieldust S, Segal I, Schechtman E, Granot I. Local injury to the endometrium doubles the incidence of successful pregnancies in patients undergoing in vitro fertilization. Fertil Steril. 2003 Jun;79(6):1317-22. doi: 10.1016/s0015-0282(03)00345-5. PMID 12798877